CLINICAL TRIAL: NCT03012711
Title: The Effectiveness of Neuromuscular Exercise Training on Core Stability and Hip Strength in Healthy Adolescent Females
Brief Title: The Effects of Neuromuscular Exercise Training on Core Stability and Hip Strength in Healthy Adolescent Females
Acronym: NME hip/core
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Jason Peeler, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS20283 (B2016:110)
Record Dates: First submitted 2016-12-15; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): Neuromuscular exercise training group will complete a 5 week NME training program
  Interventions: Other: Neuromuscular exercise training
- Control (No Intervention): Control group will have 5 weeks with no intervention prior to being re-tested

INTERVENTIONS:
Other: Neuromuscular exercise training
  Arms: Training

SUMMARY:
This study is an evaluation of the effects of a Neuromuscular training program on hip strength and core stability. It is a randomized clinical trial evaluating pre and post scores.

ELIGIBILITY:
Inclusion Criteria:

* healthy adolescent females between 12 and 18 years old

Exclusion Criteria:

* lower body injuries in the last 6 months or lower body injuries that they are currently receiving treatment
* inability to participate in 5 week NME training program

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Hip Strength - Hand Held Dynamometry | up to 6 weeks

SECONDARY OUTCOMES:
Core Stability - Dynamic Stability Sit test | up to 6 weeks